CLINICAL TRIAL: NCT04716647
Title: A Community-Based Participatory Research to Assess the Feasibility of Ayurveda Intervention in Patients With Mild-to-Moderate COVID-19
Brief Title: Feasibility of Ayurveda in Patients With Mild-to-Moderate COVID-19: A Community-Based Participatory Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Collaborators: University of Warwick (Other); Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AU/2187
Record Dates: First submitted 2021-01-18; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: Ayurveda Intervention, Community Based Participatory Research
MeSH Terms: conditions — COVID-19 | interventions — Medicine, Ayurvedic

STUDY DESIGN:
Intervention Model Description: Community Based Participatory Research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ayurveda Intervention (Experimental): Ashwagandha, Giloy and Tulsi were given in tablet form for oral administration.
  Interventions: Other: Ayurveda

INTERVENTIONS:
Other: Ayurveda — Dosage was used in common range (Ashwagandha: Doses range from 250 mg to 5 g; Giloy: range from 500mg to 1g; Tulsi: 500mg-1g) Dosage were altered based on age, weight and severity of symptoms.

SUMMARY:
Innovative strategies are required to manage COVID-19 in the communities. Back to Roots community based project was a collaborative, pilot intervention program in British Asian community to assess the efficacy and safety of Ayurveda intervention in relieving symptoms of mild-to-moderate COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* With SARS-CoV-2 infection confirmed through reverse transcription followed by polymerase chain reaction (RT- PCR),
* With mild or moderate manifestations of COVID-19
* Willing to participate, and consent by signing the informed consent and
* not involved in another clinical trial during the study

Exclusion Criteria:

* Patients suffering from severe COVID-19 Disease as per World Health Organisation criteria (REF)
* Any of the known COVID-19 complications and emergency procedures which may require shift/admission in hospital for oxygen support or intensive care unit
* Patients with ongoing immunosuppressive therapy for any reasons
* Active cancer diagnosis, on palliative treatment or requiring current therapy with antimetabolic agents, immunotherapy or radiotherapy.
* Pregnancy and lactation
* Ayurveda practitioner decision that involvement in the study is not in the patient's best interest

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Time to clinical recovery | Up to 14-days
  To evaluate the therapeutic efficacy, mean days for clinical recovery were recorded from AiM Covid Application
Proportion of patient with negative conversion in nasopharyngeal swab | Up to 14 days
  To evaluate the therapeutic efficacy, promotion of patients were recorded through AiM Covid application

SECONDARY OUTCOMES:
Clinical Outcome | Up to 14-days
  Clinical Outcome was recorded on 7-pont ordinal scale of COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, Study Director — Aarogyam UK; Dipa Modi, Study Chair — East Park Medical Centre, NHS trust, Leicester; Vishwesh Kulkarni, Principal Investigator — University of Warwick; Abhimanyu Kumar, Study Director — Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University
Locations (1):
- Aarogyam UK, Leicester, Leicestershire, United Kingdom